CLINICAL TRIAL: NCT04417582
Title: Evaluation of Life Style Modification Medical and Surgical Treatment Modalities in Patients With Obesity: An Observational Study
Brief Title: Life Style Modification Medical and Surgical Management in Patients With Obesity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2019.948
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Obesity; Weight Change, Body; Obesity; Endocrine; Obesity, Metabolically Benign
Keywords: obesity; weight loss
MeSH Terms: conditions — Obesity; Body Weight Changes; Obesity, Metabolically Benign; Weight Loss | interventions — Orlistat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- life syte modification only: obese patients followed with life style modification
  Interventions: Procedure: bariatric surgey
- medical teatment with antiobesity drugs: patients prescribed antiobesity drugs
  Interventions: Procedure: bariatric surgey
- bariatric surgery: patients undergone bariatric surgery

INTERVENTIONS:
Procedure: bariatric surgey — patients undergone bariatric surgery or prescribed antiobesity drugs
  Other Names: antiobesity drugs ,liraglutide or orlistat
  Groups: life syte modification only; medical teatment with antiobesity drugs

SUMMARY:
In this is an observational study, obese patients that administed and followed in endocrinology clinic of Marmara University Medical school hospital will follow for clinical and laboratory parameters prospectively for 5 years

DETAILED DESCRIPTION:
Following available clinical and laboratory parameters will be collected for 5 years Treatment modalities ( life stye modification, medication, bariatric surgery) eating habits quality of life body mass index , blood pressure body fat distribution (impedance measurement) laboratory parameters (serum glucose, OGTT, insülin, lipids,creatinin ,ALT AST,CBC, ferritin calcium, phosphate, Parathormone,25 OH vitamin D, vitamin B12 ,uric acid, albumin, FSH LH testosteron, estrogen ) muscle strength (dynomometer measurement) skin glikolization autoflouresent measurement Bone mineral density mesurements (femur, spine ,forarm)

ELIGIBILITY:
Inclusion Criteria:

Body mass index over 30 kg/m2 age between 18-65 years

Exclusion Criteria:

active malignancy pregnancy during involvement period chronic inflamatuar diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: obese patients refered to our tertiary center for obesity evaluation or treatment
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
weight loss | 6 months interval
  %5-10 weight loss
metabolic improvement | 6 months interval
  blood glucose
metabolic improvement | 6 month
  serum lipid levels

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Medical School Section of Endocrinology and Metabolism, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
data will be shared at the second year of recruitment